CLINICAL TRIAL: NCT03060863
Title: Targeting Self-Regulation to Promote Adherence and Health Behaviors in Children
Brief Title: ABC Brain Games Self-Regulation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alison Miller, Associate Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HUM00104622
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Self-Regulation
Keywords: children
MeSH Terms: conditions — Obesity; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1. Comparison (No Intervention): Families in this group will not receive any of the interventions.
- 2. Executive functioning (Experimental): Children in this arm will have the opportunity to use a computer-based working memory training game to practice recalling stimuli with an increasing number of presentations prior ("n-back" task).
  Interventions: Behavioral: 2. Executive Functioning
- 3. Food Bias (Experimental): Children in this arm will use a computer-based approach avoidance task to reduce attentional biases for food by using a joystick to push away images of nonhealthy foods and pull closer images of healthy foods.
  Interventions: Behavioral: 3. Food Bias
- 4. Emotion Regulation (Experimental): Children in this arm will use a computer-based, game-like relaxation training to teach emotion regulation and coping strategies.
  Interventions: Behavioral: 4. Emotion Regulation
- 5. Future orientation (Experimental): Children in this arm will participate in an interview training protocol to promote their capacity to utilize and articulate a future oriented perspective.
  Interventions: Behavioral: 5. Future orientation

INTERVENTIONS:
Behavioral: 2. Executive Functioning — Interventions will occur in 3 biweekly visits plus technology-based practice. The investigators will use computer-based working memory training to improve Executive Functioning (EF) and will use a working memory training game that has been used with children this age (N-back task).
  Arms: 2. Executive functioning
Behavioral: 3. Food Bias — The investigators will use attention-bias retraining techniques that have been tested in adults that have children practice approach and avoidance attentional strategies using a joystick and food images (healthy and unhealthy foods). Interventions will occur in 3 biweekly visits. Children in this arm will use a computer-based approach avoidance task to reduce attentional biases for food by using a joystick to push away images of nonhealthy foods and pull closer images of healthy foods.
  Arms: 3. Food Bias
Behavioral: 4. Emotion Regulation — Interventions will occur in 3 biweekly visits plus home practice. The investigators will use assisted relaxation training where children are trained to monitor and control their heart rate and skin conductance using biofeedback in a computer-game context (Journey to Wild Divine).
  Arms: 4. Emotion Regulation
Behavioral: 5. Future orientation — Interventions will occur in 3 biweekly visits. Children will participate in an interview protocol designed to enhance their capacity to visualize upcoming future events and describe them in detail, with the goal to make the "future" become "present".
  Arms: 5. Future orientation

SUMMARY:
The goal of this project is to measure childhood self-regulation targets known to be associated with obesity risk and poor adherence to medical regimens and to assess whether intervening on these mechanisms can improve self-regulation. The investigators will do so in a pre-existing cohort of low-income school-age children.

DETAILED DESCRIPTION:
Poor self-regulation (i.e., inability to harness cognitive, emotional or motivational resources to achieve goals) contributes to a number of unhealthy behaviors across the life course, including overeating, a lack of physical activity, smoking, alcoholism and substance abuse that are linked to poor long-term health. The self-regulation processes that generate the desire for such substances or that make it difficult to engage in healthy habits are theorized to begin very early in the lifespan. Targeting early self-regulation profiles that signal risk for engaging in unhealthy behaviors would allow more effective intervention. The investigators will assess self-regulation during pre-adolescence, a critical transition when children gain responsibility for managing their health choices and self-regulation becomes increasingly associated with health outcomes. Obesity is a complex health issue with early-emerging biological and behavioral precursors that are related to self-regulation; as such it is a good model for understanding a broad range of health conditions that require active self-management. Childhood obesity is also an ongoing public health crisis, with almost 25% of children overweight by age 4 years (35% by school-age). The goal of this study is to measure childhood self-regulation targets known to be associated with obesity risk and poor adherence to medical regimens and to assess whether intervening on these mechanisms can improve self-regulation. The investigators will do so in a cohort of children with a high rate of obesity who have been extensively phenotyped for bio-behavioral self-regulation and obesity risk factors from early childhood.

The aim is to, in low-income school-age children from extant cohorts, develop and field-test interventions designed to address self-regulation targets using a Multiphase Optimization Strategy (MOST) design to detect intervention effectiveness and child or family factors (e.g., maternal education, family stress, early childhood eating or stress regulation pattern) that may moderate intervention effects. The investigators hypothesize that our interventions will cause change in the self-regulation targets most closely related to the intervention components (e.g., EF-focused intervention will change EF targets).

ELIGIBILITY:
Inclusion Criteria:

* Participant in the ABC (Appetite, Behavior, and Cortisol) cohort being followed longitudinally since recruitment in 2009-2013
* Primary caregiver (mostly mother) has < 4-year college degree at time of initial enrollment (first study wave; child age ~4 years)
* Child born at 36+ weeks gestation
* Child had no significant perinatal complications.

Exclusion Criteria:

* History of food allergies or medical problems affecting growth
* Non-fluency in English
* Foster child
* Medications affecting cortisol
* Significant developmental delay.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Working Memory | 6 weeks
  Working memory is assessed using a standardized digit span task from the Wechsler Intelligence Scale for Children-WISC-IV, which requires participants to recite digits they have just heard in progressively longer sequences. The longest correct span of digits the participants repeats is the index of working memory.
Change in Inhibitory Control | 6 weeks
  Inhibitory control is measured using a go/no-go task. In this task, children are taught to play a computer-based "Zoo" game wherein their goal is to help the zookeeper find animals that have escaped and are loose in the zoo. Children are instructed to press a key to respond as fast as possible when they see the "go" stimulus (i.e., an orangutan who is "helping" the zookeeper retrieve the escaped animals, presented for 300 ms) but not when they see the no-go stimulus (i.e., any other animal that has "escaped"). The task thus requires children to demonstrate the capacity to inhibit the response to "go" when they see the "helper" animal, and indexes inhibitory control. Scores on this task are scored based on accuracy and reaction time.
Change in Behavior Rating Inventory of Executive Functioning (BRIEF) | 6 weeks
  Parents complete the 86-item Behavior Rating Inventory of Executive Function (BRIEF). The BRIEF yields two broad subscales of Behavioral Regulation and Metacognition that reflect the child's planning and organizing capabilities, attention shifting, working memory, and emotional control.
Change in emotional and behavioral displays indicating frustration | 6 weeks
  Child emotional and behavioral displays indicating frustration in response to a task designed to be frustrating (a lockbox with a wrong key) are videotaped and coded for latency to and intensity of child negative affect (e.g., frown, cry) or behavioral indicators of frustration (e.g., loud sigh, set keys down roughly).
Change in SIDES Affect dysregulation scale | 6 weeks
  Individual interview using SIDES Affect dysregulation scale to assess the child's ability to control feelings and how much strong feelings get in the way of doing things (e.g., "small problems got me very upset").
Change in Children's Emotion Management Scales | 6 weeks
  Children report on their tendency to engage in reappraisal and suppression emotion regulation strategies using the Children's Emotion Management Scales (e.g., "when I am feeling mad, I can stop myself from losing my temper"). Children report on the use of such strategies for feelings of anger, sadness, and worry and subscales are created to generate effective emotion management strategy scores for each emotion, and overall.
Change in NIH Toolbox scale | 6 weeks
  Parents report on child perceived stress responses, or how well the parent views the child's capacity to cope with stress, using the parent-report NIH Toolbox scale to assess perceived stress.
Change in Positive and Negative Affect Schedule for children | 6 weeks
  Parents report on child positive and negative mood using the Positive and Negative Affect Schedule for children, which presents parents with different positively- and negatively-valenced words and asks them to indicate which words best describe the way they perceive the child to feel, in general (e.g., upset, scared vs. interested, excited). Responses are summed to generate positive and negative affect scores.
Change in episodic future thinking | 6 weeks
  The interviewer asks children to think of three different upcoming future events that could happen over the next few days, next week, and the next few months, and to describe each event. The interview is audiotaped and later coded using an adaptation of prior coding systems.Indicators of episodic future thinking include use of rich, descriptive detail, vivid imagery, future-oriented language (e.g., "we will…"), and coherent narratives. Coding of the interviews is thus based on the level of detailed description of specific events; child use of future-oriented language; mental state language; and narrative coherence, and scores for richness of episodic future thinking language are generated.
Change in NIH Self-Efficacy | 6 weeks
  The NIH Self-Efficacy questionnaire assesses a participant's belief in his/her capacity to manage and have control over meaningful events (e.g., "I can manage to solve difficult problems if I try hard enough").
Change in Future Time Perspective subscale from the Zimbardo Time Perspective Questionnaire | 6 weeks
  Children indicate how much different items reflect their views ("I can manage to solve difficult problems if I try hard enough"; "I finish projects on time by working on them a little bit every day") and scores are generated to reflect the level of future-oriented time perspective .
Change in Ratio Reinforcing Computer Task | 6 weeks
  Relative reinforcing value (RRV) for food is determined by measuring child responses on a Ratio Reinforcing Computer Task to obtain palatable food. The child is shown how to play the game on a computer and told to play the game to win candy prizes (chocolate, gummy candy, etc.). Each computer screen displays three boxes containing different shapes, and each time a key is pressed the shapes rotate and change. When all shapes match, the child receives a point and for every five points, is given a ticket to use to redeem for candy at the end of the visit. The schedule of reinforcement begins at 10 presses to earn one point and doubles each time a ticket is earned (Progressive Ratio (PR) 20, PR 40, PR 80, PR 160, PR 320, PR 640, PR 1280, PR 2560, PR 5120, PR 10240). Food reinforcement is identified by the highest reinforcement schedule completed by the child to earn candy, with higher values indicating greater motivation to work for food, indexing food reward.
Change in implicit food bias | 6 weeks
  This task assesses implicit associations between images of chocolate and "stopping" versus "going". Children are first shown how to press buttons based on whether they see a "stop" (e.g., hand signaling stop) or a "go" signal (e.g., walk sign; 16 trials). In block 2 (48 trials) children sort the "stop" or "go" signals by pressing one of the buttons when one of the signals is paired with an image of chocolate (e.g., "go+chocolate") and the other button for the other (unpaired) signal ("stop"). In block 3 (48 trials), the pattern is reversed and children sort the "stop" or "go" signals based on the alternate signal-chocolate pairing (e.g., "stop+chocolate" vs. "go"). Scores are calculated using the D600 scoring protocol such that higher values on the task indicate a stronger implicit association between chocolate and "go" compared to chocolate and "stop" signals, suggesting an implicit bias toward chocolate.
Change in Power of Food Scale | 6 weeks
  Children complete this 15-item scale that assesses individual differences in sensitivity to food cues in the environment (e.g.. "I think about food even when I'm not truly hungry ") and the ability of these cues to increase desire for food (e.g., "If I see or smell a food I like, I get a powerful urge to have some ").

CONTACTS AND LOCATIONS:
Overall Officials: Alison Miller, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo SL, Gearhardt AN, Fredericks EM, Katz B, Sturza J, Kaciroti N, Gonzalez R, Hunter CM, Sonneville K, Chaudhry K, Lumeng JC, Miller AL. Targeted self-regulation interventions in low-income children: Clinical trial results and implications for health behavior change. J Exp Child Psychol. 2021 Aug;208:105157. doi: 10.1016/j.jecp.2021.105157. Epub 2021 Apr 25. PMID 33910138
- [Derived] Miller AL, Gearhardt AN, Fredericks EM, Katz B, Shapiro LF, Holden K, Kaciroti N, Gonzalez R, Hunter C, Lumeng JC. Targeting self-regulation to promote health behaviors in children. Behav Res Ther. 2018 Feb;101:71-81. doi: 10.1016/j.brat.2017.09.008. Epub 2017 Sep 28. PMID 29050636